CLINICAL TRIAL: NCT01014403
Title: The Delayed vs Early Enoxaparin Prophylaxis (DEEP) Study After Traumatic Brain Injury: A Randomized, Double-Blinded, Placebo Controlled Pilot Trial
Brief Title: Delayed Versus Early Enoxaparin Prophylaxis After Traumatic Brain Injury (TBI)
Acronym: DEEP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 082009-026
Record Dates: First submitted 2009-11-13; First posted 2009-11-17 (Estimated); Results first posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-12

CONDITIONS: Venous Thromboembolism; Traumatic Brain Injury
Keywords: venous thromboembolism; enoxaparin; traumatic brain injury; Venous thromboembolism prophylaxis traumatic brain injury
MeSH Terms: conditions — Venous Thromboembolism; Brain Injuries, Traumatic | interventions — Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- enoxaparin 30 mg SQ q12 hours (Experimental): Enoxaparin started at 24 hours post-injury and continued until 96 hours post-injury.
  Interventions: Drug: enoxaparin
- placebo (Placebo Comparator): vehicle administered sq q 12 hours
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: enoxaparin — Enoxaparin 30 mg sq q 12 hours
  Arms: enoxaparin 30 mg SQ q12 hours
Drug: placebo — vehicle
  Arms: placebo

SUMMARY:
Brain injured patients are at high risk for forming blood clots in the legs and lungs. For non-brain injured trauma patients, we decrease the chances of these blood clots forming by placing the patients on a low dose of the blood thinner enoxaparin. Starting patients with a brain injury on the blood thinner is problematic, however, as this can theoretically cause the brain injury to worsen. Trauma surgeons wait a variable period of time before starting this blood thinner because waiting too long can result in the formation of these blood clots in the legs and lungs. Previous research has shown that some brain injuries which are of lower severity can have enoxaparin started at 24 hours after injury if the brain injury is stable on a repeated computed tomography (CT) scan of the head. This is a pilot study designed to look at the rates of worsening of brain injury if the low dose blood thinner is started at 24 versus 96 hours post-injury.

DETAILED DESCRIPTION:
We propose to conduct a placebo-controlled non-inferiority pilot study to evaluate the rate of worsening of intracranial injury patterns after initiation of enoxaparin in TBI patients. Patient enrollment will occur at ETMC, blinded re-reading of CTs will occur at PMH, and administrative/analytical support will occur at UTSW. The study design will be a double-blind, randomized controlled trial in the ETMC Surgical Intensive Care Unit (SICU) consisting of 40 patients per arm. The decision for 80 patients was resource-based, as this is a pilot study. Further, we anticipate the need to contact 3 patients in order to obtain 1 successful recruitment.

Each arm will consist of low-risk TBI patients (defined as patients with a subdural or epidural hematoma < 8mm, intraparenchymal contusion < 2 cm, and/or single contusion per lobe) who have had a CT scan of the head without contrast at 24 hours post-injury which documents a stable injury pattern. The severity of neurologic deficit will have no bearing on their suitability for participation, and will not be considered in inclusion/exclusion criteria. After documentation of a stable intracranial injury pattern at this time interval, patients will be randomized to receive either enoxaparin 30 mg SQ every 12 hours or placebo with each regimen being initiated at 24 hours post-injury. A follow-up CT scan of the brain without contrast will be obtained on all patients 48 hours post-injury (and 24 hours after the initiation of enoxaparin/placebo). An additional CT scan of the brain without contrast will be obtained on any patient who experiences an abrupt change in neurologic exam at any time between the initiation of enoxaparin/placebo and the end of the study's interventional period at 96 hours post-injury (this time frame was chosen as it is the earliest time point at which there is universal agreement among both of our group's practitioners that enoxaparin use is safe from the risks of TBI expansion). Any patient with a worsened CT scan will have their investigational treatment discontinued at that time. At 96 hours post-injury, the interventional portion of the study will end, data collection for the primary endpoint will cease, and all patients will be placed on enoxaparin for the remainder of their hospital stay as per local standards of care. Patient participation in the study will last from the time of injury to 96 hours post-injury for the interventional part of the study, and from 96 hours post-injury until discharge from ETMC for the observational portion. While this latter time frame is obviously extremely variable, it averages approximately one to two weeks. During both the interventional and observational time periods, patients will have Duplex ultrasonography of the lower extremities performed for an edematous extremity, CT-angiography of the chest for unexplained hypoxia or tachycardia, and ventilation-perfusion scanning for suspicion of PE in the presence of a contraindication to IV contrast.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients admitted to the ETMC SICU with TBI who speak English or Spanish.

Exclusion Criteria:

1. Epidural or subdural hematoma > 8mm.
2. Intraparenchymal contusion >2 cm
3. Multiple contusions w/in one lobe
4. Subarachnoid hemorrhage in basilar or supracellar cistern and positive CTA
5. Increased TBI on 24 hr post-injury CT
6. Spinal canal hematoma
7. Nonoperative mgmt of American Association for the Surgery of Trauma (AAST) Grade IV or higher organ injury
8. Gastrointestinal hemorrhage
9. Ongoing bleeding from a pelvic fracture
10. Anticipated open reduction of long bone or pelvic fracture within study period.
11. Intracranial pressure (ICP) >20 mmHg
12. Coagulopathy consisting of International Normalized Ratio (INR)>1.5 or platelet count <50,000
13. Expect brain death/discharge in 48 hrs
14. Pre-existing dialysis dependence
15. Documented DVT at time of admission
16. Prisoners
17. Pregnancy
18. Age <18 years
19. Terminally ill patients
20. Anticoagulant use at time of injury
21. Inability to gain consent from patient or legal next-of-kin in instance of TBI, intoxication, or psychiatric diagnoses
22. Documented history of heparin allergy
23. Initial head CT >6 hours post-injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herb A Phelan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - UT-Southwestern Medical Center, Dallas, Texas
  - East Texas Medical Center, Tyler, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enoxaparin 30 mg SQ q12 Hours | Placebo
Started | 34 | 28
Completed | 34 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enoxaparin 30 mg SQ q12 Hours | Placebo | Total
Number analyzed (Participants) | 34 | 28 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (19) | 42 (17) | 41 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 22 | 16 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Worsening TBI Hemorrhage
Description: Worsening of TBI hemorrhage pattern on any scheduled or PRN CT scans after the initiation of treatment
Time Frame: 24 hours after the start of treatment/48 hours after the time of injury
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enoxaparin 30 mg SQ q12 Hours | Placebo
Number analyzed (Participants) | 34 | 28
percentage of participants | 5.9 [0.7 to 19.7] | 3.6 [0.1 to 18.3]

2. Secondary Outcome: Extracranial Hemorrhagic Complications
Description: percentage of participants that have extracranial hemorrhagic complications
Time Frame: prior to discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Enoxaparin 30 mg SQ q12 Hours | Placebo
Number analyzed (Participants) | 34 | 28
Participants | 0 | 0

3. Secondary Outcome: Count of Participants With Deep Vein Thrombosis (DVT) or Pulmonary Embolism (PE)
Time Frame: prior to discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Enoxaparin 30 mg SQ q12 Hours | Placebo
Number analyzed (Participants) | 34 | 28
Participants | 0 | 1

ADVERSE EVENTS:
Arm/Group | Enoxaparin 30 mg SQ q12 Hours | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/28
Other Adverse Events (participants affected / at risk) | 0/34 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes